CLINICAL TRIAL: NCT00320697
Title: A Trial of the Effects of Bupropion, Nicotine Replacement Therapy and CBT on Smoking Cessation and Smoking Relapse in Patients With Schizophrenia
Brief Title: Smoking Relapse Prevention in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Suffolk Mental Health Association (Other)
Responsible Party: Principal Investigator, A. Eden Evins, Director Center for Addiction Medicine, North Suffolk Mental Health Association
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CORRC 15-2005; HRC#2005-p-001950
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Smokers
Keywords: schizophrenia; smoking cessation; relapse prevention; nicotine; bupropion; cognitive behavioral therapy; nicotine replacement therapy
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Smoking Cessation | interventions — Bupropion; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Bupropion + Nicotine patch + Nicotine gum or lozenges (Other): Open label phase All enrolled subjects received weekly CBT group sessions, bupropion 300 mg/daily (if medically eligible), nicotine patch 21 mg/day, and up to 20 mg/day of nicotine gum or lozenge for prn use. Subjects set a quit date between weeks 3 and 4; a ½ hour individual CBT session to help prepare them for the quit date. The open phase groups consisted of 8 weekly CBT meetings.
  Interventions: Drug: bupropion + nicotine patch + nicotine gum or lozenges
- Bupropion + Nicotine Patch (Active Comparator): Randomized phase: Subjects who achieved 2 weeks continuous abstinence at the end of the open intervention and who are medically eligible for bupropion were eligible for the double blind, relapse prevention trial.Subjects eligible for bupropion were randomized to receive either nicotine patch and bupropion or placebo patch and pill added to CBT for 44 weeks.
  Interventions: Drug: bupropion + nicotine patch + nicotine gum or lozenges
- Placebo pill + placebo patch (Placebo Comparator): Randomized phase: Subjects who achieved 2 weeks continuous abstinence at the end of the open intervention and who are medically eligible for bupropion were eligible for the double blind, relapse prevention trial. Subjects eligible for bupropion were randomized to receive either nicotine patch and bupropion or placebo patch and pill added to CBT for 44 weeks.
  Interventions: Drug: Placebo pill + placebo patch

INTERVENTIONS:
Drug: bupropion + nicotine patch + nicotine gum or lozenges — Subjects eligible for bupropion were randomized to receive either nicotine patch and bupropion or placebo patch and pill added to CBT for 44 weeks.
  Arms: Bupropion + Nicotine Patch; Bupropion + Nicotine patch + Nicotine gum or lozenges
Drug: Placebo pill + placebo patch — Subjects eligible for bupropion were randomized to receive either nicotine patch and bupropion or placebo patch and pill added to CBT for 44 weeks.
  Arms: Placebo pill + placebo patch

SUMMARY:
This study seeks to determine if continued treatment with bupropion and nicotine replacement therapy (NRT) can reduce the smoking relapse rate in patients with schizophrenia.

DETAILED DESCRIPTION:
Background and Preliminary Data:

Between 72% and 90% of patients with schizophrenia smoke cigarettes, and schizophrenia patients are more likely than the general population to smoke and to smoke heavily (1-6). Compared with the general population, patients with schizophrenia have low smoking cessation rates, even through they can be both highly motivated and persistent in their attempts to quit smoking (7-10) and can tolerate short-term tobacco abstinence without significant exacerbation in clinical or cognitive symptoms (11, 12). Nicotine replacement therapy (NRT) and bupropion are each well tolerated by patients with schizophrenia, and bupropion is superior to placebo for smoking cessation in this population when added to CBT (13-20). However, abstinence rates have been low (4-19%) at 3-6 month follow up, whereas placebo plus CBT has produced cessation rates of 0-6%.

It has been estimated that 45% of cigarettes sold in the US are sold to people with a mental illness (21) and that in the UK and Ireland, patients with schizophrenia spend approximately one third of their weekly income on cigarettes (22, 23). Age-adjusted mortality from smoking-related diseases such as pulmonary and cardiovascular disease are two to six times higher among people with schizophrenia compared to age matched samples (24-27). More effective pharmacologic treatments for smoking cessation in patients with schizophrenia are thus urgently needed.

Combination treatment with bupropion and NRT has shown promise. In a large study in a non-psychiatric population, a combination of bupropion SR and NRT was superior to placebo and to NRT alone but not to bupropion alone for smoking cessation (28). In an open, non-randomized smoking cessation study in 115 nicotine dependent patients with co-morbid psychiatric and substance use disorders, patients treated with bupropion SR plus NRT and weekly CBT had significantly greater reduction in smoking than those on bupropion SR plus CBT, NRT plus CBT or CBT alone (29). Subjects on a combination of bupropion SR plus NRT also had significantly greater retention in the smoking cessation program and tolerated the combination treatment well.

These findings were extended to patients with schizophrenia in a 12-week, randomized, double-blind trial of bupropion or placebo added to NRT + CBT (30). In this trial, bupropion 300 mg/d or identical placebo was added to NRT and CBT for 12 weeks. NRT was given, starting on the quit date at week 4, as nicotine patch 21 mg/d for 4 weeks, 14 mg/d for 2 weeks and 7 mg/d for 2 weeks combined with nicotine gum up to 18 mg per day prn. Combination treatment with bupropion and NRT was well tolerated and more beneficial than NRT alone for significant smoking reduction in patients with schizophrenia (Table 1 & Figure 1). The combination treatment was also superior for continuous abstinence until week 8 when the dose of NRT was reduced. When subjects were taking bupropion 300 mg per day, nicotine patch 21 mg per day and prn nicotine gum up to 18 mg per day, they had a cessation rate of 52%. See Table 1. Patients began to relapse to smoking after the dose of nicotine patch was reduced to 14 mg per day and continued to relapse through the 12 month follow up.

It is our hypothesis that the 8-12 week treatment model that has been traditionally used for smoking cessation treatment is not of adequate duration for patients with schizophrenia. In our trial of bupropion combined with NRT, subjects experienced a 30% relapse rate during the taper of NRT patch from 21 mg/day to 7 mg/day while still on bupropion. In patients who are able to achieve abstinence with short-term treatment, a trial of longer duration treatment with bupropion + combination NRT at the dose used to quit smoking is warranted. It is our hypothesis that the rate of relapse to smoking will be lower with longer duration of the pharmacologic treatment used to quit smoking. Longer duration treatment can be justified in patients with schizophrenia for several reasons. First, schizophrenia patients have known abnormalities in nicotinic receptor expression and function and may benefit more than the general population from continued pharmacotherapy for maintenance of abstinence (32-34). Nicotinic receptors are reduced in number in patients with schizophrenia (32, 35) and heavy smoking in schizophrenia may be attributable to attempts to overcome a deficit in nicotinic activity. Benefits of nicotine to patients with schizophrenia include reversal of some of the specific cognitive deficits associated with schizophrenia and antipsychotic medications (36-40). Nicotine has been shown to improve learning, visual and spatial working memory, attention, auditory sensory gating smooth pursuit eye movements and reaction time (41, 42). The positive effects of chronic nicotine treatment appear to persist over time, and in some studies, improvements in cognition with chronic nicotine treatment become more robust over time (43). Secondly, the burden of morbidity and mortality of smoking related illness is high in schizophrenia such that it warrants a harm reduction approach. Continued NRT may be considered a harm reduction approach if it is associated with long term tobacco abstinence. For schizophrenia patients who are heavily addicted to tobacco products and would like to try to quit smoking, it may be appropriate to test whether higher abstinence rates can be sustained with longer-term treatment with bupropion and NRT, combined with a behavioral intervention. This study seeks to determine if continued treatment with bupropion and NRT can reduce the relapse rate in patients with schizophrenia.

Study Design:

We propose a study that will determine if continued treatment with bupropion and NRT can reduce smoking relapse rates in schizophrenia. This study has been designed with 3 phases: an initial open, 8 week smoking cessation phase, followed by a 44 week, randomized, placebo controlled, relapse prevention phase and then a 3 month follow-up phase.

One hundred and thirty adults with a diagnosis of schizophrenia or schizoaffective disorder will be entered into an 8-week open smoking cessation trial. Subjects will receive weekly cognitive behavioral therapy (CBT), bupropion 300 mg/d nicotine patch 21mg/day and up to 20 mg/day of either nicotine gum or lozenge for prn use. Those who attain abstinence and agree to participate in the relapse prevention phase(n=60-70), will be randomized, according to a double-blind, parallel group design, to receive continued treatment with a 21 mg nicotine patch and bupropion SR 300 mg or placebo added to CBT for 44 weeks. Adverse events will be documented at each visit. Study medication will be distributed bi-weekly during the double blind phase.

Study Procedures:

Baseline Measures and Screening:

1. Review of medical chart to confirm DSMIV diagnosis of schizophrenia/schizoaffective disorder and medication
2. Demographic Questionnaire
3. Clinical Rating Scales: SANS (Schedule for assessment of Negative symptoms), BPRS (Brief Psychiatric Rating Scale), Hamilton Calgary depression scale, AIMS (Abnormal Involuntary Movement Scale), SAS (Simpson Angus Scale), BAS (Barnes Akathisia Scale), Tiffany Questionnaire of Smoking Urges, State-Trait Anxiety Inventory, Snaith Hamilton Anhedonia scale, Barrett Impulsiveness Scale, SF-12 smoking Self Efficacy Questionnaire and the Wisconsin Smoking Withdrawal Scale.
4. Drug, alcohol and smoking history including Fagerstrom Test for Nicotine Dependence.
5. Cognitive tests including AX-Continuous Performance Test, WMS-III spatial span, Brief visuospatial memory test, Emotional Stroop, finger tapping, signal detection (reward responsivity) and WTAR IQ.6. Measure of reward responsivity using a signal detection test7. Expired air CO, Salivary Cotinine

8. Weight, height, pulse, blood pressure, and the UKU self-report of adverse events form.

9. Salivary Drug test to exclude current abuse of PCP, cannabis, alcohol, cocaine, methamphetamine and opiates.

10. Phlebotomy to measure metabolic health, cotinine, bupropion medication levels, genes for nicotine metabolism, and genes associated with smoking cessation and nicotine dependence. Additional serum will be stored. If there is a significant effect of continued treatment on smoking relapse, this serum will be tested for comparison of lipids and inflammatory biomarkers between groups.

1. Open Phase:

   All enrolled subjects will receive weekly CBT group sessions, bupropion 300 mg/ daily, nicotine patch 21 mg/day, and up to 20 mg/day of nicotine gum, lozenge, or nasal spray for prn use. Subjects will set a quit date between group sessions 3 and 4. The open phase groups will consist of 8 weekly CBT meetings with up to 10 participants. Subjects who achieve 2 weeks continuous abstinence at the end of the open intervention will be eligible for the double blind, relapse prevention trial.
2. Relapse Prevention Phase:

   Subjects will be randomized to receive either nicotine patch and bupropion or placebo patch and pill added to CBT for 44 weeks. Randomization will take place using a computer-generated table of random numbers.

   Visits will then take place bi-weekly for the first 4 visits then monthly throughout the relapse prevention phase for CBT group treatment. Study medication will be distributed at each visit. Smoking status will be determined at each visit with self-report and expired air CO. Medication side effects will also be recorded at each visit.
3. Follow- up Phase:

During medication taper and after medication is discontinued, subjects will attend 4 follow up visits over the next 3 months.

Clinical status using rating scales will be evaluated at visits 1, 11, 17, 20, 30 and 34. Serum levels of psychiatric medications and metabolic markers will also be monitored.

Subjects will be paid $5 for each of the group meetings during the open and relapse prevention phases. Subjects will also be paid an additional $5 for each follow-up visit they attend for self-report and $20 for clinical and cognitive assessments. Subjects who complete visits 30 and 34 at the end of the study will receive an additional $50 bonus.

Subject Selection and Recruitment:

Subjects are 130 adult outpatients with schizophrenia or schizoaffective disorder who smoke more than 10 cigarettes per day and wish to stop smoking. Subjects will be recruited by referral from treatment staff at Freedom Trail Clinic in Boston and by self-referral by responding to posted fliers in clinic waiting rooms. The Freedom Trail Clinic has established procedures for identifying and recruiting subjects for research. Clinicians and members of research teams meet each week to discuss current projects. Using this information clinicians approach their patients if they are likely to be suitable and interested in the study. Those who contact research staff about the study will be given information by a research assistant. Those who remain interested and express a desire to quit smoking will meet with a research psychiatrist. At this meeting subjects will be given further information about the study including risks and benefits and screening for eligibility criteria.

Case managers, primary care physicians and residential treatment staff within the Boston Area will also refer subjects. Research staff will meet with local case managers, residential staff and primary care physicians to inform them of the study, eligibility criteria and means of referral. Fliers will also be placed in local mental health facilities.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men aged 18-70 with DSM-IV diagnosis of schizophrenia or schizoaffective disorder by diagnostic interview and chart review.
2. Clinically stable on a stable dose of antipsychotic medication for at least one month, no current active suicidal ideation.
3. Expired air CO > 10ppm and self report of smoking >9 cigarettes per day.
4. Willing to set a smoking quit date within 3 weeks of beginning treatment.
5. Not treated with investigational medication in the past 30 days.
6. Competent to provide informed consent or able to provide assent accompanying informed consent from legal guardian.
7. Meets DSM-IV criteria for Nicotine Dependence.
8. Women of childbearing age must have a negative pregnancy test at screening and agree to use an approved form of contraception throughout the study.

Exclusion Criteria

1. Diagnosis of dementia, neurodegenerative disease, seizure disorder, current anorexia/bulimia nervosa, current substance abuse or dependence disorders, including alcohol, active within the last 3 months or any Axis I DSM-IV diagnosis other than schizophrenia or schizoaffective disorder. (*Note: Subjects with a seizure disorder who would not be medically eligible for bupropion may be allowed to participate, but will not be prescribed bupropion or randomized; rather, they will continue to receive open treatment through the relapse prevention phase.)
2. Severe or unstable angina; myocardial infarction in the past 2 weeks; untreated peptic ulcer; life-threatening arrhythmia; poorly controlled insulin dependent diabetes mellitus, uncontrolled hypertension, cerebrovascular event within six months; or allergy to nicotine patch. Serious illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic disease that is not stabilized such that hospitalization for treatment of that illness is likely within the next two months.
3. Patients who, in the investigator's opinion, pose a current severe homicide or suicide risk.
4. Subjects with a history of skin diseases (e.g. psoriasis), skin allergies, or strong reactions to topical preparations, medical dressings or tapes.
5. History of multiple head injuries with neurological sequelae or a single severe head injury with lasting neurological sequelae.
6. Treatment with doses of Clozapine> 500 mg per day without anticonvulsants.
7. Treatment with monoamine oxidase inhibitors.
8. Plan to continue to use tobacco products other than cigarettes.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness of 44 weeks extended duration combination treatment with bupropion SR and NRT compared with placebo on 7-day point-prevalence abstinence at the end of the 44-week of the randomized phase | 7-day point-prevalence abstinence at the end of the 44-week of the randomized phase

SECONDARY OUTCOMES:
To establish the safety and tolerability of bupropion SR, 300 mg/day, nicotine patch, 21 mg/day when combined with antipsychotic medications for 12 months in recently abstinent smokers with clinically stable schizophrenia | thought study completion

CONTACTS AND LOCATIONS:
Overall Officials: A Eden Evins, MD, MPH, Principal Investigator — North Suffolk Mental Health Association
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States